CLINICAL TRIAL: NCT02041390
Title: Effect of Short Message Service Intervention on Stent Removal/Exchange Adherence in Patients With Benign Pancreaticobiliary Diseases: a Prospectively Randomized, Controlled Study
Brief Title: Effect of Short Message Service Intervention on Stent Removal/Exchange Adherence in Patients With Benign Pancreaticobiliary Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20120920-5; 20120920-5 (Other: Institutional Review Board of Xijing Hospital)
Record Dates: First submitted 2014-01-18; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Short Message Service; Adherence; Stent Exchange; ERCP; Biliary Stricture

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMS group (Experimental): Patients in SMS group will receive reminding by additional SMS messages monthly after stent implantation.
  Interventions: Other: SMS reminder; Other: Conventional reminder
- Conventional reminder group (Active Comparator): Patients in control group will not receive additional SMS reminder monthly after stent implantation.
  Interventions: Other: Conventional reminder

INTERVENTIONS:
Other: SMS reminder — Each month after stent implantation, one investigator sent a text massage by SMS to inform patients the necessity of regular stent removal/exchange and the disadvantage of delayed management, and to remind them the appropriate date back to the hospital for stent management. Patients were requested to response by SMS and were encouraged to contact with the investigator if they had any questions about stent management.
  Arms: SMS group
Other: Conventional reminder — After stent implantation, all patients received oral instruction about further management. If single or multiple plastic stents were inserted, patients were informed back to our hospital at 3 months for stent removal/exchange; if FCSEMS was inserted, they were informed back to the hospital at 6 months.

SUMMARY:
Endoscopic implantation of plastic or covered metal stents is widely used in a variety of benign pancreaticobiliary diseases, including duct stricture, large or difficult stones, bile or pancreatic juice leak, etc. There are some late-stage adverse events after stent insertion, such as stent occlusion, proximal or distal migration, secondary duct injury and failure of stent removal, etc. The longer the stents were inserted, more likely the adverse events would happen.

Although the optimal time of stent placement has not been well established, it has been recommended that plastic stent should be removed/exchanged within 3-4 months and covered metal stent be removed within 6 months. However, it was not uncommon that patients with stent implantation did not follow the recommendation of further stent management by endoscopists.

Many methods have been used to improve the adherence of patients in medical service. With the advance of mobile technology and popular use of mobile phones, it was believed that the patient-centered outcome could be improved by mobile telecommunication with the timely support of a patient by a health professional. Thus we hypothesize that mobile technology, reminding the patients the necessity of stent management in time by short message service (SMS), might increase the patient adherence in patients with benign pancreaticobiliary diseases after ERCP.

ELIGIBILITY:
Inclusion Criteria:

* patients more than 18 years old with plastic or covered stent implantation for the drainage of bile or pancreatic juice.

Exclusion Criteria:

* primary or secondary sclerosing cholangitis;
* malignant or suspected malignant stricture of biliary or pancreatic duct;
* implantation of pancreatic duct stent for prevention of post-ERCP pancreatitis;
* expected survival time less than 6 months;
* plan of surgery within 6 months;
* pregnant or lactating women;
* patients who could not give informed consent.

Ages: 80 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Adherence rate of biliary stent removal/exchange | up to 1 year
  Percentage of patients adherence to stent removal/exchange within appropriate time (4 months for plastic stent or 7 months for covered stent).

SECONDARY OUTCOMES:
Stent-related adverse events | up to 1 year
  Percentage of patients with stent-related adverse events, including cholangitis, stent migration and abdominal pain, during follow.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Tuvignon N, Liguory C, Ponchon T, Meduri B, Fritsch J, Sahel J, Boyer J, Legoux JL, Escourrou J, Boustiere C, Arpurt JP, Barthet M, Tuvignon P, Bommelaer G, Ducot B, Prat F. Long-term follow-up after biliary stent placement for postcholecystectomy bile duct strictures: a multicenter study. Endoscopy. 2011 Mar;43(3):208-16. doi: 10.1055/s-0030-1256106. Epub 2011 Mar 1. PMID 21365514
- [Background] ASGE Technology Assessment Committee; Pfau PR, Pleskow DK, Banerjee S, Barth BA, Bhat YM, Desilets DJ, Gottlieb KT, Maple JT, Siddiqui UD, Tokar JL, Wang A, Song LM, Rodriguez SA. Pancreatic and biliary stents. Gastrointest Endosc. 2013 Mar;77(3):319-27. doi: 10.1016/j.gie.2012.09.026. PMID 23410693
- [Background] Kasher JA, Corasanti JG, Tarnasky PR, McHenry L, Fogel E, Cunningham J. A multicenter analysis of safety and outcome of removal of a fully covered self-expandable metal stent during ERCP. Gastrointest Endosc. 2011 Jun;73(6):1292-7. doi: 10.1016/j.gie.2011.01.043. Epub 2011 Apr 5. PMID 21470603
- [Background] Lester RT, Ritvo P, Mills EJ, Kariri A, Karanja S, Chung MH, Jack W, Habyarimana J, Sadatsafavi M, Najafzadeh M, Marra CA, Estambale B, Ngugi E, Ball TB, Thabane L, Gelmon LJ, Kimani J, Ackers M, Plummer FA. Effects of a mobile phone short message service on antiretroviral treatment adherence in Kenya (WelTel Kenya1): a randomised trial. Lancet. 2010 Nov 27;376(9755):1838-45. doi: 10.1016/S0140-6736(10)61997-6. Epub 2010 Nov 9. PMID 21071074
- [Background] Liu X, Luo H, Zhang L, Leung FW, Liu Z, Wang X, Huang R, Hui N, Wu K, Fan D, Pan Y, Guo X. Telephone-based re-education on the day before colonoscopy improves the quality of bowel preparation and the polyp detection rate: a prospective, colonoscopist-blinded, randomised, controlled study. Gut. 2014 Jan;63(1):125-30. doi: 10.1136/gutjnl-2012-304292. Epub 2013 Mar 16. PMID 23503044